CLINICAL TRIAL: NCT04879381
Title: Epidemiology of Anaerobic Bacteria in Cystic Fibrosis Patients Followed by the Perharidy Cystic Fibrosis Resource and Skills Centre, Roscoff: Descriptive and Non-interventional Study
Brief Title: Epidemiology of Anaerobic Bacteria in Cystic Fibrosis Patients: Descriptive and Non-interventional Study
Acronym: ANA-MUCO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: Sponsor
Other Study IDs: ANA-MUCO ( 29BRC18.0045)
Record Dates: First submitted 2021-02-11; First posted 2021-05-10 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cystic Fibrosis patients: Sputum samples
  Interventions: Other: Sputum samples

INTERVENTIONS:
Other: Sputum samples — During consultation, one expectoration will be performed.

SUMMARY:
Recently, the respiratory microbiota characterisation of a Cystic Fibrosis (CF) patients' cohort has highlighted the potential role of anaerobes, and specially species belonging to the genus Porphyromonas, in the first P. aeruginosa colonization.

The aim of this project is to describe the bacterial anaerobic population in the respiratory microbiota of a CF cohort. At the end of this study, an inventory of the anaerobic microbiota in CF respiratory samples will be establish in relation to the patients' pulmonary function and P. aeruginosa colonization status in order to speculate about the pulmonary anaerobes roles, still unknown.

The innovative aspect of the ANA-MUCO study is the use of a specific sample kit designed for the study which allows preserving anaerobic bacteria in sputum according to the recommendations of the International Human Microbiome Standards (IHMS). Extended-culture and molecular approaches will be performed to identify and describe the anaerobic bacteria which could be involved in the pulmonary homeostasis in CF respiratory samples.

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is a lethal genetic disease whose prognostic depends on the patients' respiratory impairment. Indeed, the airways microbial chronic colonization, particularly to Pseudomonas aeruginosa, leads to infectious exacerbations and to noteworthy respiratory function impairment and represents the main cause of morbidity and mortality. Nowadays, antibiotherapy is the main therapeutic solution to thwart bacterial development and to slow respiratory function degradation. However, during the disease progression, this therapeutical approach is limited by the bacteria accommodation and antibiotic resistance development.

Thanks to the development of high-throughput sequencing methods, the respiratory microbiota of CF patients has been mainly described and points the way to new therapeutic approaches. It has been establish that, i) from an early age, the respiratory microbiota of CF children is modified in comparison with the healthy children one, ii) bacterial diversity decrease progressively throughout the disease evolution, iii) anaerobes represent an important part of the healthy and CF respiratory microbiota. Thus pulmonary microbiota composition could be a better disease progression indicator than the only detection of P. aeruginosa in CF respiratory samples. Furthermore, the respiratory microbiota could influence the pathogenesis through direct interactions between micro-organism/micro-organism or micro-organism/host. Recently, thanks to the respiratory microbiota characterisation of a CF patients' cohort (MUCOBIOME study, 2012-2015), the potential role of anaerobes (and particularly species belonging to the genus Porphyromonas) in the first P. aeruginosa colonization has been highlighted. Indeed, the respiratory microbiota study of 34 CF patients has revealed that if patients are deprived or lowly colonized by Porphyromonas spp., the relative risk of P. aeruginosa colonization is 3.7 fold higher. Conversely, the relative abundance's increase of Porphyromonas spp. in CF patients receiving Ivacaftor treatment is correlated with the respiratory function improvement. Thus, in addition to be used as biomarker, the investigators speculate on the fact that some strict anaerobic species, such as Porphyromonas spp., could act as CF pathogens (like P. aeruginosa) competitors and limit their setting up in the airways.

The investigators see here the necessity of complementary studies in order to better characterise anaerobic bacteria in the airways. The aim of the ANA-MUCO study is to identify and describe anaerobic bacteria in sputum of a CF patients' cohort, to characterise the antibiotic resistance profiles of the anaerobic species isolated, to study the anaerobes repartition within the CF population and to evaluate the interactions between anaerobes and CF pathogens (P. aeruginosa, S. aureus, H. influenzae, …). In order to be the most exhaustive as possible in the anaerobes description, the innovative aspect of this study is the conception and the use of a specific sample kit which preserves anaerobic conditions in sputum according to the recommendations of the International Human Microbiome Standards (IHMS). Then, extended-culture and molecular approaches will be performed to identify the anaerobic bacteria which could be involved in the pulmonary homeostasis in CF respiratory samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of Cystic Fibrosis regardless of CFTR genotype
* Persons affiliated to the social security system
* Minor or major patients able to expectorate spontaneously or after induction
* Consent signed by the patient or the holder of parental authority for the children

Exclusion Criteria:

* Persons deprived of liberty, persons under guardianship or curatorship, persons in emergency situations
* Persons non affiliated to a social security system or not entitled
* Pulmonary transplant patients
* Refusal to participate to the study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Cystic Fibrosis patients
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Presence of anaerobic bacteria in sputum by culture and molecular approaches | Inclusion ( Day 0)
  The presence of anaerobic bacteria will be evaluated by culture and molecular approaches with regard of the number of sputum collected.

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève HERY-ARNAUD, Professor, Principal Investigator — University Hospital, Brest
Locations (2):
- France (2):
  - CHRU de Brest, Brest
  - Fondation Ildys, Roscoff

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Background] Nixon GM, Armstrong DS, Carzino R, Carlin JB, Olinsky A, Robertson CF, Grimwood K. Clinical outcome after early Pseudomonas aeruginosa infection in cystic fibrosis. J Pediatr. 2001 May;138(5):699-704. doi: 10.1067/mpd.2001.112897. PMID 11343046
- [Background] Cox MJ, Allgaier M, Taylor B, Baek MS, Huang YJ, Daly RA, Karaoz U, Andersen GL, Brown R, Fujimura KE, Wu B, Tran D, Koff J, Kleinhenz ME, Nielson D, Brodie EL, Lynch SV. Airway microbiota and pathogen abundance in age-stratified cystic fibrosis patients. PLoS One. 2010 Jun 23;5(6):e11044. doi: 10.1371/journal.pone.0011044. PMID 20585638
- [Background] Renwick J, McNally P, John B, DeSantis T, Linnane B, Murphy P; SHIELD CF. The microbial community of the cystic fibrosis airway is disrupted in early life. PLoS One. 2014 Dec 19;9(12):e109798. doi: 10.1371/journal.pone.0109798. eCollection 2014. PMID 25526264
- [Background] Klepac-Ceraj V, Lemon KP, Martin TR, Allgaier M, Kembel SW, Knapp AA, Lory S, Brodie EL, Lynch SV, Bohannan BJ, Green JL, Maurer BA, Kolter R. Relationship between cystic fibrosis respiratory tract bacterial communities and age, genotype, antibiotics and Pseudomonas aeruginosa. Environ Microbiol. 2010 May;12(5):1293-303. doi: 10.1111/j.1462-2920.2010.02173.x. Epub 2010 Feb 23. PMID 20192960
- [Background] Sibley CD, Surette MG. The polymicrobial nature of airway infections in cystic fibrosis: Cangene Gold Medal Lecture. Can J Microbiol. 2011 Feb;57(2):69-77. doi: 10.1139/w10-105. PMID 21326348
- [Background] Bernarde C, Keravec M, Mounier J, Gouriou S, Rault G, Ferec C, Barbier G, Hery-Arnaud G. Impact of the CFTR-potentiator ivacaftor on airway microbiota in cystic fibrosis patients carrying a G551D mutation. PLoS One. 2015 Apr 8;10(4):e0124124. doi: 10.1371/journal.pone.0124124. eCollection 2015. PMID 25853698
- [Background] Guilloux CA, Lamoureux C, Hery-Arnaud G. [Anaerobic bacteria, the unknown members of the lung microbiota]. Med Sci (Paris). 2018 Mar;34(3):253-260. doi: 10.1051/medsci/20183403014. Epub 2018 Mar 16. French. PMID 29547112
- [Background] Tunney MM, Field TR, Moriarty TF, Patrick S, Doering G, Muhlebach MS, Wolfgang MC, Boucher R, Gilpin DF, McDowell A, Elborn JS. Detection of anaerobic bacteria in high numbers in sputum from patients with cystic fibrosis. Am J Respir Crit Care Med. 2008 May 1;177(9):995-1001. doi: 10.1164/rccm.200708-1151OC. Epub 2008 Feb 8. PMID 18263800
- [Background] Smyth AR, Bell SC, Bojcin S, Bryon M, Duff A, Flume P, Kashirskaya N, Munck A, Ratjen F, Schwarzenberg SJ, Sermet-Gaudelus I, Southern KW, Taccetti G, Ullrich G, Wolfe S; European Cystic Fibrosis Society. European Cystic Fibrosis Society Standards of Care: Best Practice guidelines. J Cyst Fibros. 2014 May;13 Suppl 1:S23-42. doi: 10.1016/j.jcf.2014.03.010. PMID 24856775
- [Background] Hery-Arnaud G, Nowak E, Caillon J, David V, Dirou A, Revert K, Munck MR, Frachon I, Haloun A, Horeau-Langlard D, Le Bihan J, Danner-Boucher I, Ramel S, Pelletier MP, Rosec S, Gouriou S, Poulhazan E, Payan C, Ferec C, Rault G, Le Gal G, Le Berre R. Evaluation of quantitative PCR for early diagnosis of Pseudomonas aeruginosa infection in cystic fibrosis: a prospective cohort study. Clin Microbiol Infect. 2017 Mar;23(3):203-207. doi: 10.1016/j.cmi.2016.11.016. Epub 2016 Nov 27. PMID 27903460
- [Background] Lamoureux C, Guilloux CA, Beauruelle C, Jolivet-Gougeon A, Hery-Arnaud G. Anaerobes in cystic fibrosis patients' airways. Crit Rev Microbiol. 2019 Feb;45(1):103-117. doi: 10.1080/1040841X.2018.1549019. Epub 2019 Jan 21. PMID 30663924
- [Background] Société Française de Microbiologie. REMIC, Référentiel en Microbiologie Médicale, 2 volumes. SFM, 2015. 856 p. ISBN 9782878050325.
- [Background] CA-SFM EUCAST [En ligne]. Société Française de Microbiologie, 2013 [consulté le 11 janvier 2018]. Available on: http://www.sfmmicrobiologie.org/UserFiles/files/casfm/CASFM2013vjuin.pdf
- [Background] Héry-Arnaud et al., 2017, European patent EP17306297 Methods for predicting the risk of developping pulmonary colonization/infection by Pseudomonas aeruginosa.
- [Background] Keravec M, Mounier J, Guilloux CA, Fangous MS, Mondot S, Vallet S, Gouriou S, Le Berre R, Rault G, Ferec C, Barbier G, Lepage P, Hery-Arnaud G. Porphyromonas, a potential predictive biomarker of Pseudomonas aeruginosa pulmonary infection in cystic fibrosis. BMJ Open Respir Res. 2019 Mar 12;6(1):e000374. doi: 10.1136/bmjresp-2018-000374. eCollection 2019. PMID 30956802